CLINICAL TRIAL: NCT07207330
Title: Stroke Code: an Observational Cross-sectional Trial in Hospitals From Villavicencio, Colombia
Brief Title: Stroke Code in Hospitals From Villavicencio, Colombia
Acronym: SHIVC
Status: Recruiting | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other); Clinica Primavera (Unknown)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, ICU chief of staff, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2025_01_Stroke
Record Dates: First submitted 2025-09-01; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Ischemic Stroke
Keywords: Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Registries of patients admitted to the emergency room with stroke suspicion by neurological deficit or headache.

SUMMARY:
This is a descriptive cross-sectional study to evaluate stroke events in a hospital in the Orinoco region. It is based on reviewing a database obtained by routinely uploading patient information. The registry is designed to follow up on the activation of a stroke code for clinical purposes and as an internal communication strategy. All registries are reviewed monthly in a scientific committee to improve quality of healthcare, standardize therapeutic strategies, and optimize outcomes. The review of the registries will allow to recognize patterns of care, delays in treatment, and define adherence to guidelines.

DETAILED DESCRIPTION:
Background: Data banks or stroke registries are collected in several countries worldwide, generating information that improves patient healthcare quality.

Aim: The study aims to describe the stroke registry of patients admitted to a high-median-complexity institution.

Methodology: We wil perform a cross-sectional trial. Demographic and disease data, as well as discharge outcomes, are systematically collected in the RES-Q database. The records from the study period will be downloaded in Excel for evaluation. Numeric variables were assessed in their central distribution and dispersion, while categorical variables were presented in frequency and proportion.

Reports of stroke events in Latin America are scarce, and none were from the Colombian Orinoco region, even though there are multiple publications in the scientific literature about the use of clinical registries for stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Clinical diagnosis of stroke
* CT findings compatible with a stroke

Exclusion Criteria:

* Trauma

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admited to the emergency room
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Functional condition | 30 days
  Modified Rankin in 3 or below

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Study Chair — Hospital Departamental de Villavicencio
Locations (1):
- Clinica Primavera, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
The data contains personal information of patients restricted to hospital officials.

REFERENCES:
- [Result] Lou M, Ding J, Hu B, Zhang Y, Li H, Tan Z, Wan Y, Xu AD; Chinese Stroke Association Stroke Council Guideline Writing Committee. Chinese Stroke Association guidelines for clinical management of cerebrovascular disorders: executive summary and 2019 update on organizational stroke management. Stroke Vasc Neurol. 2020 Sep;5(3):260-269. doi: 10.1136/svn-2020-000355. Epub 2020 Jul 8. PMID 32641444
- [Result] Dhand A, Reeves MJ, Mu Y, Rosner BA, Rothfeld-Wehrwein ZR, Nieves A, Dhongade VA, Jarman M, Bergmark RW, Semco RS, Ader J, Marshall BDL, Goedel WC, Fonarow GC, Smith EE, Saver JL, Schwamm LH, Sheth KN. Mapping the Ecological Terrain of Stroke Prehospital Delay: A Nationwide Registry Study. Stroke. 2024 Jun;55(6):1507-1516. doi: 10.1161/STROKEAHA.123.045521. Epub 2024 May 24. PMID 38787926
- [Result] Fasugba O, Sedani R, Mikulik R, Dale S, Varecha M, Coughlan K, McElduff B, McInnes E, Hladikova S, Cadilhac DA, Middleton S. How registry data are used to inform activities for stroke care quality improvement across 55 countries: A cross-sectional survey of Registry of Stroke Care Quality (RES-Q) hospitals. Eur J Neurol. 2024 Jan;31(1):e16024. doi: 10.1111/ene.16024. Epub 2023 Aug 21. PMID 37540834
- [Result] Gimenez-Munoz A, Ara JR, Abad Diez JM, Campello Morer I, Perez Trullen JM. Trends in stroke hospitalisation rates and in-hospital mortality in Aragon, 1998-2010. Neurologia (Engl Ed). 2018 May;33(4):224-232. doi: 10.1016/j.nrl.2016.06.013. Epub 2016 Aug 21. English, Spanish. PMID 27554162
- [Result] Posadas-Martinez ML, Vicens J, Dawidowski AR, Martinez Von Scheidt MA, Pagotto VL, Blugerman GA, Schpilberg MG, Gadano AC. The role of registries in improving health and bridging healthcare, research, education, innovation and development: a research department perspective. J Int Med Res. 2024 Mar;52(3):3000605241233140. doi: 10.1177/03000605241233140. PMID 38460545
- [Result] Matuja SS, Ngimbwa J, Andrew L, Shindika J, Nchasi G, Kasala A, Paul IK, Ndalahwa M, Mawazo A, Kalokola F, Ngoya P, Rudovick L, Kilonzo S, Wajanga B, Massaga F, Kalluvya SE, Munseri P, Mnacho MA, Okeng'o K, Kimambo H, Manji M, Ruggajo P, Nagu T, Ahmed RA, Sheriff F, Mahawish K, Mangat H, Nguyen-Huynh MN, Saylor D, Peck R. Stroke characteristics and outcomes in urban Tanzania: Data from the Prospective Lake Zone Stroke Registry. Int J Stroke. 2024 Jun;19(5):536-546. doi: 10.1177/17474930231219584. Epub 2023 Dec 16. PMID 38031727